CLINICAL TRIAL: NCT05173675
Title: Empathy in Action: Sunshine Calls for Life With Diabetes
Acronym: EIA-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Lone Star Circle of Care (Unknown)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001571
Record Dates: First submitted 2021-12-02; First posted 2021-12-30 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes; Mental Health; Health Behavior
Keywords: Telephone; Empathy; Layperson; Self-Management; Incentives
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Psychological Well-Being; Health Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, stratified by PHQ-9 baseline scores (cut-off ≥5), on a 1:1 ratio
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research staff responsible for biomedical data collection at the sites are blinded to the status of the participant as part of control or intervention group. Self-reported outcomes are reported by participants on a tablet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program arm (Experimental): Usual Care+
  Phase 1 (6 months, months 1-6), Program. Includes empathetic communications (phone & letter), health-promoting incentives, educational materials.
  Phase 2 (6 months, months 7-12) No Program. During this follow-up period they will receive monthly SMS texts with customized messages encouraging health promoting behaviors.
  Interventions: Behavioral: Empathy in Action for life with diabetes.
- Control arm (Other): Usual Care+
  Phase 1 (6 months, months 1-6), No Program.
  Phase 2 (6 months, months 7-12) Material components of program including health-promoting incentives and educational materials.
  Interventions: Behavioral: Control Phase 2 Materials Only

INTERVENTIONS:
Behavioral: Empathy in Action for life with diabetes. — In Phase 1 (Months 1-6) participants receive ("Program"):
  1. Empathetic communications: A dedicated partner (lightly-trained lay person) who communicates with them via phone with timing and frequency defined by the participant within certain parameters. Two letters mailed during the 6 months that compile anonymized learnings from all participants in the callers panel of 10-20 participants, written as a newsletter to share back with the participant.
  2. Material Incentives: One choice of health tool (weight scale or pedometer) selected with the caller in week 1 and expected to be received in weeks 3-5. Two small recognition gifts (valued at US$25) chosen by the caller based on their understanding of the participants preferences, and sent at month 2.5 and 4.5.
  3. Educational Materials: Printed DM management educational materials mailed right after enrollment and randomization, and expected to be received in weeks 1-2.
  Arms: Program arm
Behavioral: Control Phase 2 Materials Only — 1. Material Incentives:
     a. Choice of health tool (weight scale or pedometer) and 2 health promoting gifts chosen by the caller at the end of their 6 month measurement visit.
     i. Health tool is mailed out within the 7th month ii. Health promoting gifts are mailed out in the 8th and 10th month
  2. Educational Materials a. The same educational materials mailed to participants in the intervention arm "Program" will be mailed to control arm participants after they complete their 6 months visit
  Arms: Control arm

SUMMARY:
Randomized controlled trial of the effectiveness in managing diabetes and improving mental health through a telephonic layperson-delivered empathy and relationship-focused program for patients at a Federally Qualified Health Center (FQHC) against usual care.

DETAILED DESCRIPTION:
In this study, we will assess the effectiveness of a 6-month program delivered by phone by lightly-trained lay people to individuals with diabetes, with the goal of empathetic relationship building and engagement to support day-to-day challenges of managing diabetes and working towards self-management goals. We will recruit from a collaborating Federally Qualified Health Center (FQHC) and use a randomized controlled trial, comparing program to usual care. Telephone callers will be lay people (no formal health training) who will be recruited for authentic interest and empathetic skills and lightly trained on conversational skills, cultural nuances, and how best to support people's individual lifestyle goals on nutrition, exercise, sleep and medication adherence. Callers will encourage participants to seek additional help from their clinic or specific social services as needs arise that benefit from early escalation.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≥ 7.5% at baseline measurement and 8.0% at least one time 12 months prior to study enrollment.
* At least one visit with Lone Star Circle of Care within the past 12 months (in person or telehealth)
* Willing to answer the PHQ-9 form in its entirety at baseline data collection (due to stratified randomization design).

Exclusion Criteria:

* HbA1c < 7.5% at baseline measurement.
* Refusal to answer the PHQ-9 form in its entirety at baseline data collection.
* Moderate to severe cognitive impairment
* Currently pregnant (if of female sex)
* Undergoing cancer treatment
* Having diagnosis of end-stage renal disease or serious mental illness
* Having moderate to severe cognitive impairment
* Receiving systemic treatment with prednisone or immunosuppressant therapy following an organ transplant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1c) | 6 months
  Finger stick point-of-care portable device

SECONDARY OUTCOMES:
Depression as measured by scores on the Patient Health Questionnaire 9-item (PHQ-9) | 6 months
  Self-administered. Based on the nine DSM-V criteria listed under criterion A for Major Depressive Disorder. Responders are asked to rate the frequency of depression symptoms in the last 2 weeks on a Likert scale ranging from 0 (not at all) to 3 (Nearly every day). Items are summed to provide a total score (0-27). The total score serves as a marker of severity and distress (5-9 minimal depressive symptoms; 10-14 minor depression or dysthymia; 15-27 major depressive symptoms).
Diastolic and systolic blood pressure (mmHg) | 6 months
  Direct measurement with automatic blood pressure cuff
Anxiety as measured by scores on the Generalized Anxiety Disorder 7-item (GAD-7) | 6 months
  Self-administered. Based on some of the DSM-V criteria for General Anxiety Disorder to identify probable cases of GAD along with measuring anxiety symptom severity. Responders are asked to rate the frequency of anxiety symptoms in the last 2 weeks on a Likert scale ranging from 0 (not at all) to 3 (nearly every day). Items are summed to provide a total score (0-21) to inform severity (1-4 minimal symptoms; 5-9 mild symptoms; 10-14 moderate symptoms; 15-21 severe symptoms).
General health/quality of life as measured by scores on the MOS Short-form 12-item (SF-12) | 6 months
  Self-administered. Measures physical and mental health status. Summary scores range from 0-100, with higher scores indicating a better self-reported level of health.
Medication adherence as measured by scores on the Medication Adherence Report Scale 5-item (MARS-5) | 6 months
  Self-administered. It asks respondents to rate the frequency with which the five different medication-taking behaviors occur. Each items is scored on a five-point scale (5 = never, 4 = rarely, 3 = sometimes, 2 = often, 1 = very often), with higher scores indicating higher reported adherence.
Perceived Diabetes Self-Management Scale (PDSMS) | 6 months
  Self-administered. The responses for the 8 items PDSMS items range from 1 = "Strongly Disagree" to 5 = "Strongly Agree." The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Diabetes Self-Efficacy measured by scores on the Stanford Self-Efficacy for Diabetes Scale 8-item | 6 months
  Self-Administered. Respondents are asked to score their level of confidence (scale from 1, not at all confident, to 10, totally confident) at the present time in doing tasks related to diabetes management (e.g., diet behavior, physical activity, measuring blood glycemia and others). Higher scores indicate higher self-efficacy.
Loneliness measured by scores on the 3-item UCLA Loneliness Scale | 6 months
  Self-administered. Respondents rate each item as 'Never' , 'Rarely', 'Sometimes' or 'Often'. Scores range from 3 to 9. Higher numbers imply greater loneliness.
Diabetes distress measured by the 2-item Diabetes Distress Screening Scale | 6 months
  The DDS2 is a 2-item diabetes distress screening instrument asking respondents to rate on a 6-point scale the degree to which the following items caused distress: (1) feeling overwhelmed by the demands of living with diabetes, and (2) feeling that I am often failing with my diabetes regimen. Higher scores suggest higher diabetes distress.

CONTACTS AND LOCATIONS:
Overall Officials: Maninder Kahlon, PhD, Principal Investigator — University of Texas at Austin
Locations (9):
- United States (9):
  - Lone Star Circle of Care at Ben White Health Clinic, Austin, Texas
  - Lone Star Circle of Care at El Buen Samaritano, Austin, Texas
  - Lone Star Circle of Care at Collinfield, Austin, Texas
  - Lone Star Circle of Care at Northwest Austin, Austin, Texas
  - Lone Star Circle of Care at Bastrop, Bastrop, Texas
  - Lone Star Circle of Care at Cedar Park, Cedar Park, Texas
  - Lone Star Circle of Care at Lake Aire Medical Center, Georgetown, Texas
  - Lone Star Circle of Care at Pflugerville, Pflugerville, Texas
  - Lone Star Circle of Care at Texas A&M Health Science Center, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahlon MK, Aksan NS, Aubrey R, Clark N, Cowley-Morillo M, DuBois C, Garcia C, Guerra J, Pereira D, Sither M, Tomlinson S, Valenzuela S, Valdez MR. Glycemic Control With Layperson-Delivered Telephone Calls vs Usual Care for Patients With Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2448809. doi: 10.1001/jamanetworkopen.2024.48809. PMID 39656459

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT05173675/Prot_SAP_002.pdf
  • Informed Consent Form (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT05173675/ICF_003.pdf